CLINICAL TRIAL: NCT04588610
Title: Eating Disorders Non Otherwise Specified (EDNOS) in a Population of Subjects Consulting for Severe Obesity (BMI> 35) : Prevalence and Characterization Study
Brief Title: Severe Obesity and Eating Habits (OSCAR)
Acronym: OSCAR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Arras (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-04
Record Dates: First submitted 2020-10-02; First posted 2020-10-19 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Eating Disorders; Severe Obesity
MeSH Terms: conditions — Feeding and Eating Disorders; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In anorexia nervosa,the eating disorder (ED) is the cause of thinness. In severe obesity, the overweight is a symptom. This symptom, however, is only the consequence of possibly deregulated eating behavior. The literature, focusus a specified ED of DSM-V: Binge Eating Disorder (BED) or Binge Eating, whom estimated prevalence in the severely obese population varies from 1.4 to 49% depending on the studies. The other ED, called unspecified ED (or EDNOS for Eating Disorder Non Otherwise Specified in the English literature), are much less known.

The main objective of this study is to assess the prevalence rate of unspecified ED (EDNOS or "non-BED ED") in subjects with severe obesity (BMI> 35) consulting for medical or surgical management in a General Hospital Center CSO (Specialized Obesity Center) using an adapted version of the QEWP-R, called the QEWP-RA.

DETAILED DESCRIPTION:
When it comes to weight problems, no one today disputes with anorexia nervosa that thinness is only a symptom. Thinness is the consequence of a multifactorial food restriction, in other words the consequence of an Eating Behavior Disorder (ED). The diagnosis of anorexia nervosa is made relative to the presence of diagnostic criteria listed in the DSM-V (Diagnostic and Statistical Manual V). Everyone recognizes the need for multidisciplinary care that is not limited to the prescription of re-nutrition. Imposing an increase in energy intake has never been enough to cure patients with anorexia. The multidisciplinary support offered to these subjects also seeks to understand and treat the biopsychosocial determinants that perpetuate the mechanisms of food restriction and most of the therapeutic support is based on a psychotherapeutic, individual and / or family approach. The excess weight of subjects with severe obesity (Body Mass Index> 35) suffers from a lower etiopathogenic consideration. In obese people, excess weight is, too often, considered more as the problem to be treated than as the consequence of a more complex problem. Thus, the main therapeutic means still currently used are based on simplistic thermodynamic fundamentals and are based on an imposed food restriction (diet) or even undergone (bariatric surgery procedures).

The main objective of this study is to assess the prevalence rate of unspecified ED (EDNOS or "non-BED ED") in subjects with severe obesity (BMI> 35) consulting for medical or surgical management in a General Hospital Center CSO (Specialized Obesity Center) using an adapted version of the QEWP-R, called the QEWP-RA (questionnaire on eating and weight pattern-revised and modified).

The primary endpoint will be the prevalence rate of ED not specified in the QEWP-RA.

Prospective, single-center, non-interventional study involving the human person (Category 3 of the Jardé law).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and <or = at 65 years old;
* With severe obesity (BMI> 35);
* First consultation at the Arras Hospital Nutrition Unit.

Non inclusion Criteria:

* Patients who have already undergone a nutrition consultation at Arras hospital;
* Oligophrenic patients;
* Patients under guardianship;
* Patients who cannot read or write;
* Participation in an interventional study modifying his eating behavior;
* Person deprived of liberty;
* Person under tutorship or curatorship;
* Refusal to participate in the study;
* Opposition to data processing;
* Patient not affiliated to the social security scheme

Exclusion criteria :

none

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with severe obesity (BMI> 35) who consult for the first time to lose weight at the Arras Hospital Nutrition Unit
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-08-29 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
prevalence rate of unspecified ED (EDNOS or "non-BED") in subjects with severe obesity (BMI> 35) consulting for medical or surgical management in a hospital. CSO general hospital center (Specialized Obesity Center). | 1 jour
  The main objective of this study is to assess the prevalence rate of unspecified ED (EDNOS or "non-BED ED") in subjects with severe obesity (BMI> 35) consulting for medical or surgical management in a General Hospital Center CSO (Specialized Obesity Center) using an adapted version of the QEWP-R, called the QEWP-RA.

SECONDARY OUTCOMES:
To compare the prevalence rate of "BED" subjects obtained from 3 different questionnaires (Questionnaire on Eating and Weight Pattern-R (QEWP-R), Eating Disorder Examination-Questionnaire (EDE-Q) and the Binge Eating Scale (BES)). | 1 jour
  * The QEWP-R (used to diagnose Binge Eating Disorder / Purging Bulimia Nervosa / Nonpurging Bulimia Nervosa)
  * The EDE-Q : 28 item self-report questionnaire. It concerns behaviors over a 28-day time period and retains the scoring system of 0-6: 0 = behaviour was absent and 6 = behaviour was present daily or to an extreme degree
  * The BES is composed of 16 items corresponding to groups of sentences including one to be selected from 3 to 4 propositions, which best describe how one feels. For each item, the subject has to choose the formulation that best corresponds to his current situation, which results in a score varying between 0 and 3 or between 0 and 2 for each item. Half of the items measure eating behaviours and the other half assess feelings or cognitions occurring during compulsive episodes. It gives a total score (from 0 to 46) that reflects the severity of the BED. A score greater than or equal to 18 indicates significant bulimic hyperphagia.
To compare the psychopathological profiles of "BED" subjects and "EDNOS" subjects (comparison of averages (Hospital Anxiety and Depression scale (HADS), Dutch Eating Behaviour Questionnaire (DEBQ),Emotional Eating Scale(EES)). | 1 jour
  * The HADS consists of two parts: (a) 7 questions for screening for depression, and (b) 7 questions for screening for anxiety disorders. Each question receives a score between 0 and 3. The score for each part is obtained by adding the items that make up the part. The higher the score, the greater the severity of the corresponding symptoms.
  * The DEBQ is a 33-item self-report questionnaire to assess three distinct eating behaviors in adults: (1) emotional eating, (2) external eating, and (3) restrained eating. Items on the DEBQ range from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the eating behavior.
  * The EES Self-reported frequency of emotional eating is measured with the 25-item EES. Each item is scored on a 5-point scale ranging from 1 (no desire to eat) to 5 (overwhelming desire to eat). Total scores range from 25-125. Higher scores indicate more emotional eating.The EES Scale yields 3 subscales: anger/ Frustration, anxiety and depression.
To compare emotional eating profiles of "BED" subjects and "EDNOS" subjects (Comparison of emotional eating profiles (Hospital Anxiety and Depression scale (HADS), Dutch Eating Behaviour Questionnaire (DEBQ), Emotional Eating Scale(EES))). | 1 jour
  * The HADS consists of two parts: (a) 7 questions for screening for depression, and (b) 7 questions for screening for anxiety disorders. Each question receives a score between 0 and 3. The score for each part is obtained by adding the items that make up the part. The higher the score, the greater the severity of the corresponding symptoms.
  * The DEBQ is a 33-item self-report questionnaire to assess three distinct eating behaviors in adults: (1) emotional eating, (2) external eating, and (3) restrained eating. Items on the DEBQ range from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the eating behavior.
  * The EES Self-reported frequency of emotional eating is measured with the 25-item EES. Each item is scored on a 5-point scale ranging from 1 (no desire to eat) to 5 (overwhelming desire to eat). Total scores range from 25-125. Higher scores indicate more emotional eating.The EES Scale yields 3 subscales: anger/ Frustration, anxiety and depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Arras General Hospital, Arras, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Zwaan M. Binge eating disorder and obesity. Int J Obes Relat Metab Disord. 2001 May;25 Suppl 1:S51-5. doi: 10.1038/sj.ijo.0801699. PMID 11466589
- [Background] Hudson JI, Lalonde JK, Berry JM, Pindyck LJ, Bulik CM, Crow SJ, McElroy SL, Laird NM, Tsuang MT, Walsh BT, Rosenthal NR, Pope HG Jr. Binge-eating disorder as a distinct familial phenotype in obese individuals. Arch Gen Psychiatry. 2006 Mar;63(3):313-9. doi: 10.1001/archpsyc.63.3.313. PMID 16520437
- [Background] Gormally J, Black S, Daston S, Rardin D. The assessment of binge eating severity among obese persons. Addict Behav. 1982;7(1):47-55. doi: 10.1016/0306-4603(82)90024-7. PMID 7080884
- [Background] Yanovski SZ. Binge eating disorder: current knowledge and future directions. Obes Res. 1993 Jul;1(4):306-24. doi: 10.1002/j.1550-8528.1993.tb00626.x. PMID 16350580
- [Background] Spitzer RL, Yanovski S, Wadden T, Wing R, Marcus MD, Stunkard A, Devlin M, Mitchell J, Hasin D, Horne RL. Binge eating disorder: its further validation in a multisite study. Int J Eat Disord. 1993 Mar;13(2):137-53. PMID 8477283
- [Background] Striegel-Moore RH, Dohm FA, Solomon EE, Fairburn CG, Pike KM, Wilfley DE. Subthreshold binge eating disorder. Int J Eat Disord. 2000 Apr;27(3):270-8. doi: 10.1002/(sici)1098-108x(200004)27:33.0.co;2-1. PMID 10694712
- [Background] Striegel-Moore RH, Wilson GT, Wilfley DE, Elder KA, Brownell KD. Binge eating in an obese community sample. Int J Eat Disord. 1998 Jan;23(1):27-37. doi: 10.1002/(sici)1098-108x(199801)23:13.0.co;2-3. PMID 9429916